CLINICAL TRIAL: NCT04743934
Title: RAD 2003/XUAB2104: Randomized Phase II Trial of Flibanserin in Men Receiving Androgen Suppression for Prostate Cancer
Brief Title: Flibanserin in Men Receiving Androgen Suppression for Prostate Cancer
Acronym: RAD 2003
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew McDonald (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrew McDonald, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300006880; 5R21CA259808-02 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Prostate Adenocarcinoma
Keywords: Flibanserin; Androgen Deprivation Therapy (ADT)
MeSH Terms: interventions — flibanserin; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flibanserin + ADT (Experimental): Flibanserin at 100mg by mouth once daily at bedtime while receiving androgen deprivation therapy (ADT).
  Interventions: Drug: Flibanserin 100 MG; Drug: Androgen deprivation therapy
- Placebo + ADT (Placebo Comparator): Placebo at 100mg by mouth once daily at bedtime while receiving androgen deprivation therapy (ADT).
  Interventions: Drug: Placebo; Drug: Androgen deprivation therapy

INTERVENTIONS:
Drug: Flibanserin 100 MG — Flibanserin 100mg tablets taken by mouth daily at bedtime
  Arms: Flibanserin + ADT
Drug: Placebo — Visually identical placebo tablets taken by mouth daily at bedine
  Arms: Placebo + ADT
Drug: Androgen deprivation therapy — Androgen deprivation therapy consisting of a GnRH agonist or antagonist, choice of agent at discretion of treating physician.

SUMMARY:
This is a double-blinded, placebo-controlled randomized phase II clinical trial investigating whether flibanserin promotes sexual interest in men with prostate cancer who are receiving androgen suppression.

DETAILED DESCRIPTION:
More than 40,000 men with prostate cancer in the United States will begin androgen deprivation therapy (ADT) each year. ADT is an important part of treatment, because it improves survival for men with metastatic or high-risk localized disease, and reduces rates of biochemical progression for men with intermediate-risk localized disease who receive radiation. The most common ADT agents modulate gonadotropin-releasing hormone to suppress the downstream testosterone production, resulting in testosterone levels similar to those observed following surgical castration (<20 ng/dL). Since male sexual interest is highly correlated with serum testosterone levels, loss of sexual interest is nearly universal among men who receive ADT.Sexual dysfunction is the most common complaint among men with prostate cancer and contributes to lower overall quality of life (QoL) experienced by men receiving ADT. Furthermore, the loss of sexual interest experienced during ADT is highly distressing for men with prostate cancer and their partners, which contributes additional psychological morbidity in these patients.

Flibanserin is approved for treatment of female hypoactive sexual desire disorder, and the safety profile of 100mg daily flibanserin is well described in premenopausal women.The safety profile of flibanserin in healthy men has been assessed in multiple phase I clinical trials, but has not been evaluated among men receiving ADT for prostate cancer.

This is a phase II randomized, double-blinded, placebo-controlled clinical trial designed to provide an initial estimate of the efficacy of flibanserin to promote sexual interest in men with prostate cancer receiving androgen suppression therapy and to confirm the safety profile. This study will take place at a single academic comprehensive cancer center.

Following confirmation of eligibility, participants who are enrolled in this study are randomized to receive daily flibanserin 100mg or placebo for a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to take oral medication and be willing to adhere to the study regimen.
* Male age >18 years.
* Histologically confirmed prostate cancer.
* Currently receiving gonadotropin releasing hormone agonist/antagonist monotherapy.
* Serum testosterone <50 ng/dL.
* Serum AST and ALT less than 2 times upper limit of normal.
* Endorsed reduced sexual interest.
* Attempted intercourse.
* Current sexual partner.
* Was sexually active with partner within 6 months prior to ADT.
* No other antineoplastic therapy planned during study period.
* No active symptoms attributable to systemic prostate cancer.

Exclusion Criteria:

* Current systemic prostate cancer treatment besides GnRH agonist/antagonist, anti-androgens, or abiraterone.
* Prior to ADT had erections not firm enough for intercourse despite use of pharmacologic agents such as phosphodiesterase-5 inhibitors.
* Current symptoms attributable to active prostate cancer
* Moderate or heavy alcohol use (>2 drinks/day)
* Concurrent moderate or strong CYP3A4 inhibitors
* Concurrently taking medication classified as a monoamine oxidase inhibitor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient-reported frequency of attempting sexual intercourse | Baseline up to 12 weeks
  The number of patients in each arm reporting attempting sexual intercourse at least 3 times in the prior month (0-2 attempts vs. 3+ attempts) will be compared using the two-group chi-square test, or Fisher's exact test if the assumptions for the chi-square test are not tenable.

SECONDARY OUTCOMES:
Sexual Quality of Life (QoL) | Up to 12 weeks
  Determined using T-scores (higher T-score indicates better QoL) from the PROMIS v2.0 Brief Sexual Function and Satisfaction (Male) form and comparing T-score between patients receiving flibanserin and patients receiving placebo.
Frequency of physician-assessed grade 3+ Adverse Events | Baseline up to 12 weeks
  Toxicity will be assessed by a physician investigator and scored using the CTCAE v5.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McDonald, MD, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided